CLINICAL TRIAL: NCT03087396
Title: A Longitudinal Outcomes Study of the Subchondroplasty® Procedure in the Foot/Ankle
Status: Completed | Type: Observational
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Other Study IDs: KC.CR.I.AM.16.2
Record Dates: First submitted 2017-02-21; First posted 2017-03-22 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-01

CONDITIONS: Insufficiency Fractures; Stress Fracture; Stress Fracture, Ankle, Foot and Toes
Keywords: bone marrow defect; bone marrow lesion; stress fracture; calcium phosphate; bone substitute material
MeSH Terms: conditions — Fractures, Stress

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Treatment of insufficiency fractures — Filling of micro fractures or insufficiency fractures with a bone substitute material

SUMMARY:
Post Market clinical outcomes study to collect data on the short - and long-term outcomes for subjects who are undergoing or who have undergone the Subchondroplasty Procedure in the foot and/or ankle in a standard clinical setting. Outcomes to be assessed include pain medication usage, pain, function, activity levels and patient satisfaction.

DETAILED DESCRIPTION:
This is a post-market, multi-center, patient outcomes centered study to evaluate the on-label use of AccuFill during the Subchondroplasty procedure (SCP). Enrolled subjects will sign an informed consent form, satisfy the inclusion/exclusion criteria and have at least one bone marrow lesion, such as a cyst or stress fracture confirmed by diagnostic imaging in the foot and/or ankle joint. Demographics, medical history and medications will recorded at the time of enrollment. Surgical details including the SCP procedure, concomitant surgical procedures and intraoperative safety events will be recorded. Subjects will complete validated patient reported outcomes measures pre-operatively including the Foot Function Index (FFI) revised short form, the EQ-5D™ and numeric pain score. These measures plus a subject satisfaction survey will also be administered post-operatively at 6 weeks, 3 months, 6 months, 1 year, and 2 years. Screening for adverse events and revision surgeries will occur throughout the study.

Target enrollment is 140 patients at up to 25 clinical sites. Subjects will complete the study at 2 years or will be withdrawn if the patient undergoes revision surgery of the Subchondroplasty site.

ELIGIBILITY:
Inclusion Criteria:

* Subject has at least one bone defect such as a bone marrow lesion (BML), cyst or stress fracture confirmed by diagnostic imaging
* Surgeon considers the patient appropriate for the SCP procedure
* Subject provides voluntary signature on the Institutional Review Board (IRB) approved Informed Consent
* Subject is at least 18 years of age
* Subject must be physically and mentally willing and able, in the Investigator's opinion at the time of enrollment, to complete outcome forms via the internet, telephone or regular mail

Exclusion Criteria:

* Subject is pregnant at the time of surgery
* Subject is incarcerated
* Subject is involved in active litigation related to the condition being treated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Approximately 140 subjects, each with at least one bone marrow lesion (BML) in any of the bones of the foot and/or ankle who have elected to undergo or have undergone the Subchondroplasty (SCP) procedure will be enrolled in the study.
Sampling Method: Non-Probability Sample
Enrollment: 148 (Actual)
Dates: Start 2017-03-10 (Actual); Primary Completion 2023-08-23 (Actual); Study Completion 2023-08-23 (Actual)

PRIMARY OUTCOMES:
Change from baseline Foot Function Index-Revised (FFI-R) short form score at 12 Months | 12 months
  Change from baseline score, range 0-100, for patient reported pain, stiffness, difficulty, activity limitation and social issues at 12 months.

SECONDARY OUTCOMES:
Incidence and severity of device and/or procedure related adverse events and re-visions/re-operations | 5 years
  Summary and description of procedure and device related adverse events and surgical re-operations and relatedness to the bone substitute material and procedure
Change in numeric pain score from baseline at 12 Months | 12 months
  Change in numeric pain score using a 0-10 scale from baseline at 12 months.
Change in EuroQol-5 Dimensions (EQ-5D) from baseline at 12 months | 12 months
  Change in patient quality of life from baseline at 12 months. A scoring function is created using a population preference weighted health index. The change from the baseline score will be measured at 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Robert B Anderson, MD, Principal Investigator — OrthoCarolina Research Institute, Inc.
Locations (12):
- United States (11):
  - OrthoArizona, Mesa, Arizona
  - The CORE Institute, Sun City, Arizona
  - OrthoNorcal, Capitola, California
  - Eisenhower Desert Orthopedic Center, Rancho Mirage, California
  - Stanford University Medical Center, Orthopedics, Redwood City, California
  - University of California, Davis, Sacramento, California
  - Capital Orthopaedics and Sports Medicine, Clive, Iowa
  - Podiatry Center of the Lehigh Valley, Bethlehem, Pennsylvania
  - Rothman Institute, Bryn Mawr, Pennsylvania
  - Premier Orthopaedics & Sports Medicine, Exton, Pennsylvania
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- St. Paul's Hospital (Providence Health), Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No